CLINICAL TRIAL: NCT06847737
Title: Prediction of Hypotension After Spinal Anesthesia in Cesarean Sections Using Non-Invasive Measurement Methods: Comparative Analysis of Perfusion Index, Pulse Variability Index, Tissue Oxygen Saturation and Tissue Hemoglobin Index
Brief Title: Prediction of Hypotension After Spinal Anesthesia in Cesarean Sections Using Non-Invasive Measurement Methods
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. prof, Istinye University
Other Study IDs: haseki nırs masimo
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Postspinal Hypotension
MeSH Terms: interventions — Perfusion Index

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: perfusion index — To compare the incidence of hypotension after spinal anesthesia and the values of perfusion index, pleth variability index, tissue oxygen saturation and tissue hemoglobin index between those who developed hypotension and those who did not develop hypotension over time.
  Other Names: pleth variability index; tissue hemoglobin index; tissue oxygen saturation

SUMMARY:
To compare the incidence of hypotension after spinal anesthesia and the values of perfusion index, pleth variability index, tissue oxygen saturation and tissue hemoglobin index between those who developed hypotension and those who did not develop hypotension over time.

ELIGIBILITY:
Inclusion Criteria:

* Those who underwent elective cesarean section over the age of 18,
* American Society of Anesthesia I and II,
* Agree to participate in the study,

Exclusion Criteria:

* <18 or >45 years,
* preeclampsia,
* cardiovascular disorders,
* fetal abnormalities,
* not undergoing spinal anesthesia or undergoing general anesthesia during surgery,
* not agreeing to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women who will have a cesarean section
Study Population: Fifty pregnant women over the age of 18 who underwent elective cesarean section, were American Society of Anesthesia I and II, and agreed to participate in the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
tissue oxygen saturation | 4 month
  which indicates an increase in local tissue perfusion
tissue hemoglobin index | 4 month
  indicating vasodilation

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ilies C, Kiskalt H, Siedenhans D, Meybohm P, Steinfath M, Bein B, Hanss R. Detection of hypotension during Caesarean section with continuous non-invasive arterial pressure device or intermittent oscillometric arterial pressure measurement. Br J Anaesth. 2012 Sep;109(3):413-9. doi: 10.1093/bja/aes224. Epub 2012 Jul 12. PMID 22798273
- [Result] Kuwata S, Suehiro K, Juri T, Tsujimoto S, Mukai A, Tanaka K, Yamada T, Mori T, Nishikawa K. Pleth variability index can predict spinal anaesthesia-induced hypotension in patients undergoing caesarean delivery. Acta Anaesthesiol Scand. 2018 Jan;62(1):75-84. doi: 10.1111/aas.13012. Epub 2017 Oct 16. PMID 29034983
- [Result] Duggappa DR, Lokesh M, Dixit A, Paul R, Raghavendra Rao RS, Prabha P. Perfusion index as a predictor of hypotension following spinal anaesthesia in lower segment caesarean section. Indian J Anaesth. 2017 Aug;61(8):649-654. doi: 10.4103/ija.IJA_429_16. PMID 28890560